CLINICAL TRIAL: NCT02824432
Title: Exploratory Study of the Effect of Omega-3-acid Ethyl Esters on Vascular Endothelial Function in Patients With Hyperlipidemia by Flow Mediated Dilation
Brief Title: Exploratory Study of the Effect of Omega-3-acid Ethyl Esters (TAK-085) on Vascular Endothelial Function in Patients With Hyperlipidemia by Flow Mediated Dilation
Acronym: Oasis Flow
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: TAK-085-4001; U1111-1182-6745 (Other: WHO); JapicCTI-163269 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2016-05-20; First posted 2016-07-06 (Estimated); Results first posted 2019-05-06 (Actual); Last update posted 2019-05-06 (Actual); Status verified 2019-01

CONDITIONS: Hyperlipidemia
MeSH Terms: conditions — Hyperlipidemias | interventions — TAK-085

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAK-085 2g (Experimental): A dose of 2 grams of omega-3-acid ethyl esters (TAK-085) will be orally administered once a day immediately after meal.
  Interventions: Drug: TAK-085
- TAK-085 4g (Experimental): A dose of 4 grams of omega-3-acid ethyl esters (TAK-085) will be orally administered twice a day immediately after meal.
  Interventions: Drug: TAK-085

INTERVENTIONS:
Drug: TAK-085 — TAK-085 capsules

SUMMARY:
The purpose of this study is to explore the effects of omega-3-acid ethyl esters (TAK-085) on vascular endothelial function when administered for 8 weeks, as measured by FMD, in patients with hyperlipidemia.

DETAILED DESCRIPTION:
This is a multicenter, collaborative, randomized, open-label study designed to explore the effects of administration of omega-3-acid ethyl esters (TAK-085) [2 g (2 g PO QD) or 4 g (2 g PO BID) for 8 weeks] on vascular endothelial function, as measured by flow-mediated dilation (FMD), in patients receiving a hydroxymethylglutaryl-coenzyme A (HMG-CoA) reductase inhibitor and have concurrent hypertriglyceridemia.

Considering the potential bias by factors that affect FMD between treatment groups, stratified allocation will be performed with fasting triglyceride (TG) level as a factor.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with the diagnosis of hyperlipidemia and receiving instructions for lifestyle improvement
2. Participants with a fasting TG level of 150 -499 mg/dL at Visit 1 after informed consent (Day -29 to Day -1 before start of study drug administration)
3. Participants receiving a stable dose of HMG-CoA reductase inhibitor therapy continuously for at least 4 weeks before informed consent at Visit 1 (Day -29 to Day -1 before start of study drug administration)
4. Male or postmenopausal female participants
5. Participants who, in the opinion of the principal investigator or the investigator, are capable of understanding the content of the clinical research and complying with the research protocol requirements.
6. Participants who can provide written informed consent prior to the conduction of the clinical research procedures
7. Participants aged ≥20 years at the time of informed consent at Visit 1(Day -28 to Day 0 before the start of study drug administration)

Exclusion Criteria:

1. Participants with a history of revascularization or those have had coronary artery disease (a definitive diagnosis of myocardial infarction, angina) within 24 weeks before informed consent at Visit 1 (Day -29 to Day -1 before the start of study drug administration)
2. Participants who have undergo aortic aneurysmectomy within 24 weeks prior to informed consent at Visit 1 (Day -29 to Day -1 before the start of study drug administration) or those with concurrent aortic aneurysm
3. Participants who have had clinically significant hemorrhagic disorders (e.g., hemophilia, capillary fragility, gastrointestinal ulcer, urinary tract hemorrhage, hemoptysis, and vitreous hemorrhage) within 24 weeks prior to informed consent at Visit 1 (Day -29 to Day -1 before the start of study drug administration) or those who concurrently have the above disorders
4. Participant with a fasting FMD level of 0% measured at the start of study drug administration at Visit 2 (Day -15 to Day -1 before the start of study drug administration)
5. Participants in whom the type and dosage of HMG-CoA reductase inhibitors, antidiabetic drugs and antihypertensive drugs have been changed within 4 weeks prior to informed consent at Visit 1 (Day -29 to Day -1 before the start of study drug administration)
6. Participants who have started anti dyslipidemic agents within 4 weeks prior to informed consent at Visit 1 (Day -29 to Day -1 before the start of study drug administration)
7. Participants requiring a change in the dose of dyslipidemia therapeutic, antidiabetic, or antihypertensive drugs during the period between informed consent at Visit 1 (Day -29 to Day -1 before the start of study drug administration) and the start of study drug administration at Visit 2 (Day -15 to Day -1 before the start of study drug administration)
8. Participants with severe hepatic dysfunction
9. Participants with severe renal dysfunction (as an indicator, CKD category ≥G3b, equivalent to an A3)
10. Participants who have been diagnosed with pancreatitis
11. Participants who have been diagnosed with lipoprotein lipase deficiency, apoprotein C-II deficiency, familial hypercholesterolemia, familial combined hyperlipidemia, or familial type III hyperlipidemia
12. Participants with concurrent Cushing's syndrome, uremia, systemic lupus erythematosus (SLE), serum dysproteinemia, or hypothyroidism
13. Participants with symptomatic Peripheral Arterial Disease (PAD)
14. Participants with concurrent hypertension of grade II or higher Note 1) Note 1: Participants with systolic blood pressure of ≥160 mm Hg or diastolic BP of ≥100 mm Hg regardless of treatment with antihypertensive drugs
15. Participants who are habitual drinkers drinking an average of over 100 mL per day (expressed in terms of quantity of alcohol) or participants with, or with a history of drug abuse or addiction Note 2)
16. Participants with a history of hypersensitivity or allergy for omega-3-acid ethyl esters-
17. Participants who smoke
18. Participants participating in other clinical studies
19. Participants who have been determined to be ineligible as subjects in the study by the principal investigator or the investigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2016-08-04 (Actual); Primary Completion 2017-08-19 (Actual); Study Completion 2017-08-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (4):
- Japan (4):
  - Yufu, Oita Prefecture
  - Shinjuku, Tokyo
  - Kagoshima
  - Ōita

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available after applicable marketing approvals and commercial availability have been received, an opportunity for the primary publication of the research has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com/approach for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

REFERENCES:
- [Derived] Teramoto T, Shibata H, Suzaki Y, Matsui S, Uemura N, Tomiyama H, Yamashina A. Discrepancy Between Fasting Flow-Mediated Dilation and Parameter of Lipids in Blood: A Randomized Exploratory Study of the Effect of Omega-3 Fatty Acid Ethyl Esters on Vascular Endothelial Function in Patients With Hyperlipidemia. Adv Ther. 2020 May;37(5):2169-2183. doi: 10.1007/s12325-020-01286-1. Epub 2020 Mar 21. PMID 32200533

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 7 investigative sites in Japan, from 04 August 2016 to 19 August 2017.
Pre-assignment Details: Participants with a historical diagnosis of hyperlipidemia were enrolled in one of two groups, omega-3-acid ethyl esters (TAK-085) 2 grams (g) and TAK-085 4 g treatment groups.
Groups:
- TAK-085 2 g: A dose of 2 g of omega-3-acid ethyl esters (TAK-085) was orally administered once a day immediately after meal.
- TAK-085 4 g: A dose of 4 g of omega-3-acid ethyl esters (TAK-085) was orally administered twice a day immediately after meal.
Period: Overall Study
Arm/Group | TAK-085 2 g | TAK-085 4 g
Started | 18 | 19
Completed | 17 | 19
Not Completed | 1 | 0
Not completed — Major Protocol Deviation | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set, The safety analysis set was defined as all participants who received at least one dose of the study drug during the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | TAK-085 2 g | TAK-085 4 g | Total
Number analyzed (Participants) | 18 | 19 | 37
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.5 (11.14) | 61.5 (7.94) | 60.1 (9.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 22
  Male | 7 | 8 | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: Participants]
  Japan | 18 | 19 | 37
Height [Mean (Standard Deviation); unit: Centimeters (cm)] | 158.4 (9.08) | 162.1 (9.21) | 160.3 (9.21)
Weight [Mean (Standard Deviation); unit: Kilograms (kg)] | 68.34 (13.288) | 71.94 (14.636) | 70.19 (13.921)
BMI [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index = weight (kg)/[height (m)^2]
  kg/m^2 | 27.12 (4.097) | 27.14 (3.483) | 27.13 (3.740)
Duration of Dyslipidemia [Mean (Standard Deviation); unit: Years] — Mean duration between start of study and first time of diagnosis of dyslipidemia was reported.
  Years | 9.24 (5.924) | 9.51 (5.173) | 9.38 (5.474)
Postmenopausal Period [Mean (Standard Deviation); unit: Years] — Population: This baseline characteristic was analyzed only in female participants with available data for analysis.
  Years
    number analyzed (Participants) | 9 | 8 | 17
    (all) | 9.9 (6.11) | 16.6 (5.88) | 13.1 (6.77)
Frequency of Consumption of Fish [Count of Participants; unit: Participants] — Participants were asked a question about frequency of consumption of fish and answered from 4 types of the answers; Almost Every Day, About Every 2 Days, About Once or Twice per Week, and Rarely. Reported data were the number of participants who selected from 4 answers.
  Participants
    Almost Every Day | 1 | 1 | 2
    About Every 2 days | 5 | 2 | 7
    About Once or Twice per Week | 11 | 12 | 23
    Rarely | 1 | 4 | 5
Smoking History [Count of Participants; unit: Participants]
  Never Smoked | 13 | 9 | 22
  Ex-Smoker | 5 | 10 | 15
Drinking History [Count of Participants; unit: Participants] — Participants who answered Yes or No for a question "Drink Alcohol Almost Every Day?" were reported.
  Participants
    Yes | 4 | 2 | 6
    No | 14 | 17 | 31
Triglyceride (TG) level (fasting) [Mean (Standard Deviation); unit: Milligram (mg)/deciliter (dL)] | 176.8 (59.18) | 194.4 (48.57) | 185.8 (53.96)
TG level (4 h postprandial) [Mean (Standard Deviation); unit: mg/dL] | 265.9 (102.63) | 278.2 (70.54) | 272.2 (86.60)
EPA/AA ratio [Mean (Standard Deviation); unit: Ratio] — EPA: Eicosapentaenoic acid, AA: Arachidonic acid
  Ratio | 0.265 (0.1156) | 0.240 (0.1551) | 0.252 (0.1360)

OUTCOME MEASURES:

1. Primary Outcome: Flow-mediated Dilation (FMD) With Fasting State at Baseline, Week 4 and Week 8
Description: FMD refers to dilation (widening) of an artery when blood flow increases in that artery. To determine FMD, brachial artery dilation following a transient period of forearm ischemia is measured using ultrasound. FMD was calculated by the value of Maximum diastolic vessel size minus vessel size at rest, divided by vessel size at rest, described with percentage.
Time Frame: Prior to meal at Baseline, Week 4, and Week 8
Population: Full analysis set (FAS); FAS was defined as participants who were randomized and received at least one dose of the study drug. The number analyzed is the number of participants with data available for analysis at the given time-point.
Measure: Mean (Standard Deviation); unit: Percentage of dilation
Arm/Group | TAK-085 2 g | TAK-085 4 g
Number analyzed (Participants) | 18 | 19
Percentage of dilation
  Baseline: number analyzed (Participants) | 17 | 17
  Baseline | 6.71 (3.466) | 5.85 (3.615)
  Week 4: number analyzed (Participants) | 16 | 17
  Week 4 | 5.85 (1.920) | 3.15 (2.898)
  Week 8: number analyzed (Participants) | 16 | 17
  Week 8 | 5.38 (2.279) | 3.95 (2.244)

2. Primary Outcome: Change From Baseline in FMD With Fasting State at Week 4 and Week 8
Description: as for outcome 1
Time Frame: Prior to meal at Baseline and Week 4, and Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of dilation
Arm/Group | TAK-085 2 g | TAK-085 4 g
Number analyzed (Participants) | 18 | 19
Percentage of dilation
  Week 4: number analyzed (Participants) | 15 | 17
  Week 4 | -1.02 (2.782) | -2.71 (3.480)
  Week 8: number analyzed (Participants) | 15 | 15
  Week 8 | -1.20 (3.638) | -1.33 (2.754)

3. Primary Outcome: Percent Change From Baseline in FMD With Fasting State at Baseline, Week 4 and Week 8
Description: as for outcome 1
Time Frame: Prior to meal at Baseline and Week 4, and Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent of Change
Arm/Group | TAK-085 2 g | TAK-085 4 g
Number analyzed (Participants) | 18 | 19
Percent of Change
  Week 4: number analyzed (Participants) | 15 | 17
  Week 4 | 24.01 (143.217) | -36.70 (52.824)
  Week 8: number analyzed (Participants) | 15 | 15
  Week 8 | 37.37 (218.483) | -8.19 (52.111)

4. Secondary Outcome: FMD With 4-Hours Postprandial State at Baseline and Week 8
Description: as for outcome 1
Time Frame: 4-hours after meal at Baseline and Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of dilation
Arm/Group | TAK-085 2 g | TAK-085 4 g
Number analyzed (Participants) | 18 | 19
Percentage of dilation
  Baseline: number analyzed (Participants) | 14 | 15
  Baseline | 5.49 (2.489) | 3.80 (2.267)
  Week 8: number analyzed (Participants) | 15 | 18
  Week 8 | 5.81 (2.848) | 4.95 (2.516)

5. Secondary Outcome: Change From Baseline in FMD With 4-Hours Postprandial State at Week 8
Description: as for outcome 1
Time Frame: 4-hours after meal at Baseline and Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of dilation
Arm/Group | TAK-085 2 g | TAK-085 4 g
Number analyzed (Participants) | 13 | 15
Percentage of dilation | 0.02 (1.284) | 1.02 (3.519)

6. Secondary Outcome: Percent Change From Baseline in FMD With 4-Hours Postprandial State at Week 8
Description: as for outcome 1
Time Frame: 4-hours after meal at Baseline and Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent of Change
Arm/Group | TAK-085 2 g | TAK-085 4 g
Number analyzed (Participants) | 13 | 15
Percent of Change | -1.62 (31.542) | 76.79 (132.271)

7. Secondary Outcome: Triglyceride (TG) Level With Fasting State at Baseline, Week 4, and Week 8
Time Frame: Prior to meal at Baseline, Week 4, and Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | TAK-085 2 g | TAK-085 4 g
Number analyzed (Participants) | 18 | 19
mg/dL
  Baseline | 176.8 (59.18) | 194.4 (48.57)
  Week 4 | 178.2 (75.49) | 144.6 (39.36)
  Week 8: number analyzed (Participants) | 17 | 19
  Week 8 | 157.2 (45.80) | 144.9 (43.05)

8. Secondary Outcome: Change From Baseline in TG Level With Fasting State at Week 4 and Week 8
Time Frame: Prior to meal at Baseline and Week 4, and Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | TAK-085 2 g | TAK-085 4 g
Number analyzed (Participants) | 18 | 19
mg/dL
  Week 4 | 1.4 (69.58) | -49.8 (35.67)
  Week 8: number analyzed (Participants) | 17 | 19
  Week 8 | -23.1 (48.40) | -49.4 (46.68)

9. Secondary Outcome: Percent Change From Baseline in TG Level With Fasting State at Week 4 and Week 8
Time Frame: Prior to meal at Baseline and Week 4, and Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent of Change
Arm/Group | TAK-085 2 g | TAK-085 4 g
Number analyzed (Participants) | 18 | 19
Percent of Change
  Week 4 | 4.8 (34.17) | -24.5 (15.14)
  Week 8: number analyzed (Participants) | 17 | 19
  Week 8 | -7.7 (31.26) | -23.5 (22.12)

10. Secondary Outcome: TG Level With 4-Hours Postprandial State at Baseline, Week 4 and Week 8
Time Frame: 4-hours after meal at Baseline, Week 4, and Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | TAK-085 2 g | TAK-085 4 g
Number analyzed (Participants) | 18 | 19
mg/dL
  Baseline | 265.9 (102.63) | 278.2 (70.54)
  Week 4: number analyzed (Participants) | 17 | 19
  Week 4 | 266.1 (75.18) | 216.2 (79.11)
  Week 8: number analyzed (Participants) | 17 | 19
  Week 8 | 240.5 (74.66) | 202.3 (78.26)

11. Secondary Outcome: Change From Baseline in TG Level With 4-Hours Postprandial State at Week 4 and Week 8
Time Frame: 4-hours after meal at Baseline and Week 4, and Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | TAK-085 2 g | TAK-085 4 g
Number analyzed (Participants) | 18 | 19
mg/dL
  Week 4: number analyzed (Participants) | 17 | 19
  Week 4 | -9.1 (89.29) | -62.1 (54.28)
  Week 8: number analyzed (Participants) | 17 | 19
  Week 8 | -34.7 (89.40) | -75.9 (57.02)

12. Secondary Outcome: Percent Change From Baseline in TG Level With 4-Hours Postprandial State at Week 4 and Week 8
Time Frame: 4-hours after meal at Baseline and Week 4, and Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent of Change
Arm/Group | TAK-085 2 g | TAK-085 4 g
Number analyzed (Participants) | 18 | 19
Percent of Change
  Week 4: number analyzed (Participants) | 17 | 19
  Week 4 | 3.8 (29.15) | -22.4 (18.54)
  Week 8: number analyzed (Participants) | 17 | 19
  Week 8 | -6.0 (35.29) | -27.2 (21.09)

13. Secondary Outcome: Dihomo-gamma-linolenic Acid Concentration With Fasting State at Baseline, Week 4 and Week 8
Description: Samples for plasma fatty acid fractions (Dihomo-gamma-linolenic acid, Arachidonic acid, Eicosapentaenoic acid, Docosahexaenoic acid, EPA/AAratio, and DHA/AAratio) were taken under the fasting condition. Reported data was the observation value at each point.
Time Frame: Prior to meal at Baseline, Week 4 and Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: microgram (μg)/milliliter (mL)
Arm/Group | TAK-085 2 g | TAK-085 4 g
Number analyzed (Participants) | 18 | 19
microgram (μg)/milliliter (mL)
  Baseline | 51.37 (14.761) | 57.32 (12.274)
  Week 4 | 42.54 (11.493) | 34.37 (7.777)
  Week 8: number analyzed (Participants) | 17 | 19
  Week 8 | 43.12 (9.060) | 33.32 (8.609)

14. Secondary Outcome: Change From Baseline in Dihomo-gamma-linolenic Acid Concentration With Fasting State at Week 4 and Week 8
Description: Samples for plasma fatty acid fractions (Dihomo-gamma-linolenic acid, Arachidonic acid, Eicosapentaenoic acid, Docosahexaenoic acid, EPA/AAratio, and DHA/AAratio) were taken under the fasting condition. Reported data was the change from baseline in Dihomo-gamma-linolenic acid at each time point.
Time Frame: Prior to meal at Baseline and Week 4, and Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | TAK-085 2 g | TAK-085 4 g
Number analyzed (Participants) | 18 | 19
μg/mL
  Week 4 | -8.83 (11.838) | -22.95 (10.112)
  Week 8: number analyzed (Participants) | 17 | 19
  Week 8 | -9.91 (9.338) | -24.01 (10.093)

15. Secondary Outcome: Percent Change From Baseline in Dihomo-gamma-linolenic Acid Concentration With Fasting State at Week 4 and Week 8
Description: Samples for plasma fatty acid fractions (Dihomo-gamma-linolenic acid, Arachidonic acid, Eicosapentaenoic acid, Docosahexaenoic acid, EPA/AAratio, and DHA/AAratio) were taken under the fasting condition. Reported data was the percent change from baseline in Dihomo-gamma-linolenic acid at each time point.
Time Frame: Prior to meal at Baseline and Week 4, and Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent of Change
Arm/Group | TAK-085 2 g | TAK-085 4 g
Number analyzed (Participants) | 18 | 19
Percent of Change
  Week 4 | -12.99 (23.659) | -38.81 (12.362)
  Week 8: number analyzed (Participants) | 17 | 19
  Week 8 | -15.11 (20.541) | -41.09 (12.981)

16. Secondary Outcome: Arachidonic Acid Concentration With Fasting State at Baseline, Week 4 and Week 8
Description: as for outcome 13
Time Frame: Prior to meal at Baseline, Week 4 and Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | TAK-085 2 g | TAK-085 4 g
Number analyzed (Participants) | 18 | 19
μg/mL
  Baseline | 254.36 (52.266) | 253.08 (69.609)
  Week 4 | 238.69 (65.009) | 217.96 (49.583)
  Week 8: number analyzed (Participants) | 17 | 19
  Week 8 | 243.71 (76.318) | 197.82 (49.991)

17. Secondary Outcome: Change From Baseline in Arachidonic Acid Concentration With Fasting State at Week 4 and Week 8
Description: Samples for plasma fatty acid fractions (Dihomo-gamma-linolenic acid, Arachidonic acid, Eicosapentaenoic acid, Docosahexaenoic acid, EPA/AAratio, and DHA/AAratio) were taken under the fasting condition. Reported data was the change from baseline in Arachidonic acid at each time point.
Time Frame: Prior to meal at Baseline and Week 4, and Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | TAK-085 2 g | TAK-085 4 g
Number analyzed (Participants) | 18 | 19
μg/mL
  Week 4 | -15.67 (32.588) | -35.12 (37.533)
  Week 8: number analyzed (Participants) | 17 | 19
  Week 8 | -10.50 (39.241) | -55.26 (36.603)

18. Secondary Outcome: Percent Change From Baseline in Arachidonic Acid Concentration With Fasting State at Week 4 and Week 8
Description: Samples for plasma fatty acid fractions (Dihomo-gamma-linolenic acid, Arachidonic acid, Eicosapentaenoic acid, Docosahexaenoic acid, EPA/AAratio, and DHA/AAratio) were taken under the fasting condition. Reported data was the percent change from baseline in Arachidonic acid at each time point.
Time Frame: Prior to meal at Baseline and Week 4, and Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent of Change
Arm/Group | TAK-085 2 g | TAK-085 4 g
Number analyzed (Participants) | 18 | 19
Percent of Change
  Week 4 | -6.66 (13.212) | -11.80 (12.789)
  Week 8: number analyzed (Participants) | 17 | 19
  Week 8 | -5.41 (15.195) | -20.19 (12.200)

19. Secondary Outcome: Eicosapentaenoic Acid Concentration With Fasting State at Baseline, Week 4 and Week 8
Description: as for outcome 13
Time Frame: Prior to meal at Baseline, Week 4 and Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | TAK-085 2 g | TAK-085 4 g
Number analyzed (Participants) | 18 | 19
μg/mL
  Baseline | 66.04 (29.246) | 55.62 (26.992)
  Week 4 | 128.07 (34.223) | 192.34 (43.711)
  Week 8: number analyzed (Participants) | 17 | 19
  Week 8 | 134.94 (41.173) | 193.75 (45.718)

20. Secondary Outcome: Change From Baseline in Eicosapentaenoic Acid Concentration With Fasting State at Week 4 and Week 8
Description: Samples for plasma fatty acid fractions (Dihomo-gamma-linolenic acid, Arachidonic acid, Eicosapentaenoic acid, Docosahexaenoic acid, EPA/AAratio, and DHA/AAratio) were taken under the fasting condition. Reported data was the change from baseline in Eicosapentaenoic acid at each time point.
Time Frame: Prior to meal at Baseline and Week 4, and Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | TAK-085 2 g | TAK-085 4 g
Number analyzed (Participants) | 18 | 19
μg/mL
  Week 4 | 62.02 (36.430) | 136.72 (45.047)
  Week 8: number analyzed (Participants) | 17 | 19
  Week 8 | 70.98 (32.197) | 138.13 (53.122)

21. Secondary Outcome: Percent Change From Baseline in Eicosapentaenoic Acid Concentration With Fasting State at Week 4 and Week 8
Description: Samples for plasma fatty acid fractions (Dihomo-gamma-linolenic acid, Arachidonic acid, Eicosapentaenoic acid, Docosahexaenoic acid, EPA/AAratio, and DHA/AAratio) were taken under the fasting condition. Reported data was the percent change from baseline in Eicosapentaenoic acid at each time point.
Time Frame: Prior to meal at Baseline and Week 4, and Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent of Change
Arm/Group | TAK-085 2 g | TAK-085 4 g
Number analyzed (Participants) | 18 | 19
Percent of Change
  Week 4 | 126.17 (85.878) | 297.49 (140.921)
  Week 8: number analyzed (Participants) | 17 | 19
  Week 8 | 137.55 (94.717) | 305.92 (153.767)

22. Secondary Outcome: Docosahexaenoic Acid Concentration With Fasting State at Baseline, Week 4 and Week 8
Description: as for outcome 13
Time Frame: Prior to meal at Baseline, Week 4 and Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | TAK-085 2 g | TAK-085 4 g
Number analyzed (Participants) | 18 | 19
μg/mL
  Baseline | 173.30 (51.854) | 145.43 (45.037)
  Week 4 | 207.04 (51.493) | 212.20 (47.226)
  Week 8: number analyzed (Participants) | 17 | 19
  Week 8 | 201.04 (47.958) | 207.53 (48.728)

23. Secondary Outcome: Change From Baseline in Docosahexaenoic Acid Concentration With Fasting State at Week 4 and Week 8
Description: Samples for plasma fatty acid fractions (Dihomo-gamma-linolenic acid, Arachidonic acid, Eicosapentaenoic acid, Docosahexaenoic acid, EPA/AAratio, and DHA/AAratio) were taken under the fasting condition. Reported data was the change from baseline in Docosahexaenoic acid at each time point.
Time Frame: Prior to meal at Baseline and Week 4, and Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | TAK-085 2 g | TAK-085 4 g
Number analyzed (Participants) | 18 | 19
μg/mL
  Week 4 | 33.74 (42.605) | 66.77 (41.677)
  Week 8: number analyzed (Participants) | 17 | 19
  Week 8 | 26.31 (31.103) | 62.11 (51.694)

24. Secondary Outcome: Percent Change From Baseline in Docosahexaenoic Acid Concentration With Fasting State at Week 4 and Week 8
Description: Samples for plasma fatty acid fractions (Dihomo-gamma-linolenic acid, Arachidonic acid, Eicosapentaenoic acid, Docosahexaenoic acid, EPA/AAratio, and DHA/AAratio) were taken under the fasting condition. Reported data was the percent change from baseline in Docosahexaenoic acid at each time point.
Time Frame: Prior to meal at Baseline and Week 4, and Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent of Change
Arm/Group | TAK-085 2 g | TAK-085 4 g
Number analyzed (Participants) | 18 | 19
Percent of Change
  Week 4 | 24.32 (29.608) | 52.83 (35.072)
  Week 8: number analyzed (Participants) | 17 | 19
  Week 8 | 19.69 (26.183) | 51.54 (44.898)

25. Secondary Outcome: Eicosapentaenoic Acid to Arachidonic Acid (EPA/AA) Ratio With Fasting State at Baseline, Week 4 and Week 8
Description: Samples for plasma fatty acid fractions (Dihomo-gamma-linolenic acid, Arachidonic acid, Eicosapentaenoic acid, Docosahexaenoic acid, EPA/AAratio, and DHA/AAratio) were taken under the fasting condition.
Time Frame: Prior to meal at Baseline, Week 4 and Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | TAK-085 2 g | TAK-085 4 g
Number analyzed (Participants) | 18 | 19
Ratio
  Baseline | 0.265 (0.1156) | 0.240 (0.1551)
  Week 4 | 0.564 (0.1990) | 0.946 (0.3722)
  Week 8: number analyzed (Participants) | 17 | 19
  Week 8 | 0.579 (0.1811) | 1.043 (0.3881)

26. Secondary Outcome: Change From Baseline in EPA/AA Ratio With Fasting State at Week 4 and Week 8
Description: Samples for plasma fatty acid fractions (Dihomo-gamma-linolenic acid, Arachidonic acid, Eicosapentaenoic acid, Docosahexaenoic acid, EPA/AAratio, and DHA/AAratio) were taken under the fasting condition. Reported data was the change from baseline in EPA/AA Ratio at each time point.
Time Frame: Prior to meal at Baseline and Week 4, and Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | TAK-085 2 g | TAK-085 4 g
Number analyzed (Participants) | 18 | 19
Ratio
  Week 4 | 0.299 (0.1714) | 0.706 (0.2874)
  Week 8: number analyzed (Participants) | 17 | 19
  Week 8 | 0.322 (0.1301) | 0.803 (0.3241)

27. Secondary Outcome: Percent Change From Baseline in EPA/AA Ratio With Fasting State at Week 4 and Week 8
Description: Samples for plasma fatty acid fractions (Dihomo-gamma-linolenic acid, Arachidonic acid, Eicosapentaenoic acid, Docosahexaenoic acid, EPA/AAratio, and DHA/AAratio) were taken under the fasting condition. Reported data was the percent change from baseline in EPA/AA Ratio at each time point.
Time Frame: Prior to meal at Baseline and Week 4, and Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent of Change
Arm/Group | TAK-085 2 g | TAK-085 4 g
Number analyzed (Participants) | 18 | 19
Percent of Change
  Week 4 | 141.396 (94.4914) | 353.990 (162.5131)
  Week 8: number analyzed (Participants) | 17 | 19
  Week 8 | 152.244 (95.3802) | 412.899 (202.3624)

28. Secondary Outcome: Docosahexaenoic Acid to Arachidonic Acid (DHA/AA) Ratio With Fasting State at Baseline, Week 4 and Week 8
Description: as for outcome 25
Time Frame: Prior to meal at Baseline, Week 4 and Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | TAK-085 2 g | TAK-085 4 g
Number analyzed (Participants) | 18 | 19
Ratio
  Baseline | 0.697 (0.2163) | 0.619 (0.2795)
  Week 4 | 0.913 (0.2874) | 1.038 (0.3726)
  Week 8: number analyzed (Participants) | 17 | 19
  Week 8 | 0.881 (0.2673) | 1.119 (0.4178)

29. Secondary Outcome: Change From Baseline in DHA/AA Ratio With Fasting State at Week 4 and Week 8
Description: Samples for plasma fatty acid fractions (Dihomo-gamma-linolenic acid, Arachidonic acid, Eicosapentaenoic acid, Docosahexaenoic acid, EPA/AAratio, and DHA/AAratio) were taken under the fasting condition. Reported data was the change from baseline in DHA/AA ratio at each time point.
Time Frame: Prior to meal at Baseline and Week 4, and Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | TAK-085 2 g | TAK-085 4 g
Number analyzed (Participants) | 18 | 19
Ratio
  Week 4 | 0.216 (0.1782) | 0.419 (0.2170)
  Week 8: number analyzed (Participants) | 17 | 19
  Week 8 | 0.177 (0.1512) | 0.499 (0.3002)

30. Secondary Outcome: Percent Change From Baseline in DHA/AA Ratio With Fasting State at Week 4 and Week 8
Description: Samples for plasma fatty acid fractions (Dihomo-gamma-linolenic acid, Arachidonic acid, Eicosapentaenoic acid, Docosahexaenoic acid, EPA/AAratio, and DHA/AAratio) were taken under the fasting condition. Reported data was the percent change from baseline in DHA/AA ratio at each time point.
Time Frame: Prior to meal at Baseline and Week 4, and Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent of Change
Arm/Group | TAK-085 2 g | TAK-085 4 g
Number analyzed (Participants) | 18 | 19
Percent of Change
  Week 4 | 33.538 (27.8356) | 76.932 (52.6408)
  Week 8: number analyzed (Participants) | 17 | 19
  Week 8 | 27.797 (26.0796) | 93.582 (69.6390)

31. Secondary Outcome: Number of Participants Reporting One or More Adverse Events (AEs)
Time Frame: Up to Week 8
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | TAK-085 2 g | TAK-085 4 g
Number analyzed (Participants) | 18 | 19
Participants | 4 | 2

32. Secondary Outcome: Number of Participants Reporting One or More AEs Related to Body Weight
Time Frame: Up to Week 8
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | TAK-085 2 g | TAK-085 4 g
Number analyzed (Participants) | 18 | 19
Participants | 0 | 0

33. Secondary Outcome: Number of Participants Reporting One or More AEs Related to Blood Pressure in the Sitting Position
Time Frame: Up to Week 8
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | TAK-085 2 g | TAK-085 4 g
Number analyzed (Participants) | 18 | 19
Participants | 0 | 0

34. Secondary Outcome: Number of Participants Reporting One or More AEs Related to Pulse in the Sitting Position
Time Frame: Up to Week 8
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | TAK-085 2 g | TAK-085 4 g
Number analyzed (Participants) | 18 | 19
Participants | 0 | 0

35. Secondary Outcome: Number of Participants Reporting One or More AEs Related to Laboratory Tests of Fasting Plasma Glucose
Time Frame: Up to Week 8
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | TAK-085 2 g | TAK-085 4 g
Number analyzed (Participants) | 18 | 19
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to Week 8
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | TAK-085 2 g | TAK-085 4 g
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/19
Other Adverse Events (participants affected / at risk) | 4/18 | 2/19
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TAK-085 2 g (N=18) | TAK-085 4 g (N=19)
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2016-07-07): https://cdn.clinicaltrials.gov/large-docs/32/NCT02824432/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-14): https://cdn.clinicaltrials.gov/large-docs/32/NCT02824432/SAP_001.pdf